CLINICAL TRIAL: NCT07189598
Title: Phase III Study of Adaptive Stereostactic Body Radiotherapy With Dose-escalation on the Dominant Intraprostatic Lesion for High-risk Prostate Cancer: ORION Trial Protocol
Brief Title: Phase III Adaptive Adaptive Stereostactic Body Radiotherapy (SBRT) With Dose Escalation for High-Risk Prostate Cancer
Acronym: ORION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2-75-001
Record Dates: First submitted 2025-09-15; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-09

CONDITIONS: High Risk Prostate Cancer
Keywords: phase III; stereotactic body radiotherapy; prostate cancer; high-risk; randomized clinical trial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- innovative arm (Experimental): Participants treated with Stereostatic Body RadioTherapy (SBRT) will be administered an adaptative stereostactic, ultra-fractionated radiotherapy every other day, for a total treatment time of 10 days. Total treatment time should not exceed 17 days
  Interventions: Procedure: Adaptive Stereostatic Body RadioTherapy (SBRT) including both Whole Pelvic RadioTherapy (WPRT) and dose-escalation on the Dominant Intraprostatic Lesion (DIL)
- control arm (Active Comparator): Patients will be treated by Conventional fractionation in 39 fractions, 5 days a week or Moderate hypofractionation in 20 fractions , 5 days a week
  Interventions: Procedure: conventional or a moderately hypofractionated

INTERVENTIONS:
Procedure: Adaptive Stereostatic Body RadioTherapy (SBRT) including both Whole Pelvic RadioTherapy (WPRT) and dose-escalation on the Dominant Intraprostatic Lesion (DIL) — The doses delivered will be:
  * the prostate gland, at a dose of 36.25 Gray, in 5 fractions,
  * the dominant intraprostatic lesion, up to 50 Gray, in 5 fractions,
  * seminal vesicles, at a dose of 25 Gray in 5 fractions,
  * pelvic lymph nodes, at 25 Gray in 5 fractions
  Arms: innovative arm
Procedure: conventional or a moderately hypofractionated — * Conventional fractionation includes the prescription of a total dose of 78 Gray in 39 fractions to the prostate gland (and seminal vesicles, in case of T3b disease), and a dose de 50Gy in 25 fractions to pelvic nodal areas.
  * Moderate hypofractionation includes the prescription of a total dose of 60 Gray to the prostate gland (and seminal vesicles, in case of T3b disease), and 44 Gray to pelvic nodal areas in 20 fractions using a simultaneous integrated boost (SIB)
  Arms: control arm

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy of adaptive prostate Stereotatic Body RadioTherapy (SBRT), which integrates both Whole Pelvic RadioTherapy (WPRT) and dose escalation on the Dominant Intraprostatic Lesion (DIL), compared with standard radiotherapy. This will be assessed using a 5-year cost-utility analysis based on data from the clinical trial and the National Health Data System (NHDS).

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Age ≥ 18 years
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Histologically proven prostate adenocarcinoma, not previously treated
* High-risk or very high-risk according to the National Comprehensive Cancer Network (NCCN) :

  * T3a / T3b (proximal extension only),
  * and/or ISUP (International Society of Urological Pathology) grade 4-5,
  * and/or PSA (Prostate-Specific Antigen) 20ng/mL
* Non-metastatic, as proven by Prostate Specific Membrane Antigen (PSMA) positron emission tomography/computed tomography (PET/CT) and pelvic MRI (Magnetic Resonance Imaging) less than 2 months before starting hormone therapy
* Normal testosterone levels prior to hormone therapy
* Ability to give consent for inclusion in the study
* Acceptance of treatment and monitoring modalities

Exclusion Criteria:

* Presence of nodal or distant metastases
* Stage T4.
* Prostate volume > 80 cm3.
* IPSS >19/35.
* Previous local treatment of prostate adenocarcinoma (HIFU (High-Intensity Focused Ultrasound), cryotherapy)
* Previous TransUrethral Resection of the prostate (PTUR)).
* Previous pelvic radiotherapy.
* Chronic inflammatory bowel disease.
* Active cardiovascular comorbidities (e.g. myocardial infarction or ischemic stroke within the last 6 months).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2032-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of adaptive prostate Stereostatic Body RadioTherapy (SBRT) integrating both Whole Pelvic RadioTherapy (WPRT) and dose-escalation on the Dominant Intraprostatic Lesion (DIL) | Five years after radiotherapy
  The primary endpoint is incremental cost effectiveness ratio (ICER) expressed as the cost for each healthy life-year gained at 5 years, with costs estimated from the National Health Data System (NHDS), overall survival (defined as the time between the 1st day of treatment and death from any cause), and utility estimated from clinical trial data

SECONDARY OUTCOMES:
Biochemical recurrence-free survival | Up to Year 5
  defined as the time between date of randomization and date of biochemical recurrence, with biological recurrence defined according to Phoenix criteria.
Metastatic recurrence-free survival | Up to Year 5
  Defined as the time from date of randomization to date of metastatic recurrence, metastatic recurrence being defined as the appearance of a lesion outside the target volume.
Overall survival | Up to Year 5
  Defined as the time from date of randomization to date of death (from any cause)
Quality of life | Up to Year 5
  defined with International Prostate Symptoms Score (IPSS)
Quality of life | Up to Year 5
  Defined with Expanded Prostate Cancer Index Composite (EPIC) score
Quality of life | Up to Year 5
  Defined with European Quality Of Life -5 Dimensions-5 Levels (EQ-5D-5L) scales
Toxicity (GenitoUrea, GenitoIntestial, sexual) of the experimental arm | Up to Year 5
  graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0